CLINICAL TRIAL: NCT06534905
Title: Pilot Randomized Controlled Trial of E-cigarette Switching Among Older Adults With Opioid Use Disorder
Brief Title: E-cigarette Switching Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Bethea A Kleykamp, Assistant Professor, University of Maryland School of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HP-00110720
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Use; Opioid Use Disorder; Tobacco-Related Disorders
Keywords: e-cigarette
MeSH Terms: conditions — Tobacco Use; Opioid-Related Disorders; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Intervention is an e-cigarette (not an FDA approved treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E-cigarette switching (Active Comparator): NJOY Ace e-cigarette (menthol or tobacco flavor, depending on patient preference) to be used ad libitum.
  Interventions: Other: E-cigarette
- Standard brief advice to address tobacco use (Other): Usual Care/Treatment As Usual Patients will be exposed to a brief smoking cessation intervention (BI) based on long-standing tobacco treatment guidelines (Fiore, 2008) and recommendations in the newly revised 4th edition of the ASAM. If a patient reports wanting to stop smoking, they will be instructed to reach out to their medical provider at the treatment clinic. They will be given multiple state and federal resources for quitting smoking.
  If the patient does not want to quit smoking during the brief intervention, we will check with them during the next session about their interest.
  The brief smoking intervention will be delivered at each session to check on individuals who are attempting to quit and to possibly motivate those who aren't quitting to initiate a quit attempt.
  Interventions: Behavioral: Control/Standard Advice

INTERVENTIONS:
Other: E-cigarette — Each participant assigned to the e-cigarette group will given a rechargeable NJOY Ace e-cigarette that is either tobacco or mint-flavored (based on their preference). Participants will also be given disposable pods prefilled with nicotine. When the pod is empty, the participant will throw it away and replace it with a new pod provided by the study staff. Participants will be asked to use as little or as much of the e-cigarette during their study participation, including choosing not to use the product. Participants will also be given information on the relative harms of nicotine and tobacco products as recommended by the American Society of Addiction Medicine.
  Other Names: ENDS; vaporized nicotine
  Arms: E-cigarette switching
Behavioral: Control/Standard Advice — Brief advice to quit according recommendations from the American Society of Addiction Medicine
  Arms: Standard brief advice to address tobacco use

SUMMARY:
The goal of this clinical trial is to learn if adults 50 years and older who currently smoke tobacco and are in treatment for opioid use disorder will switch to using e-cigarettes instead of continued smoking. Participants will not have a plan to quit smoking and will not be actively trying to quit smoking at the start of the trial. The main questions the study aims to answer are:

* Are e-cigarettes a feasible and acceptable harm-reduction tool among older adults who currently smoke tobacco and don't have a plan to quit?
* Will switching to e-cigarettes and reducing tobacco use be more likely among patients given access to e-cigarettes compared to individuals who are exposed to a standard brief intervention for smoking cessation (control)?
* Does the accuracy of nicotine/tobacco knowledge change after participants are exposed to education on the harms of nicotine relative to no education?

Participants will complete a baseline session (BL) and follow-up visits at weeks 2, 6, and 8, each lasting 30-90 minutes, for a total of approximately 3-4 hours of participation in the study. Each session will include computerized assessments of tobacco and other substance use, health status, mood, and functioning.

Patients will be randomly assigned at baseline (if meeting eligibility criteria) to receive an e-cigarette product (name of product: NJOY Ace) or brief advice to quit smoking (in alignment with recommendations by the American Society of Addiction Medicine).

DETAILED DESCRIPTION:
Volunteers will be patients diagnosed with opioid use disorder (OUD) who have been in medication-based treatment (methadone or buprenorphine) at the University of Maryland Addiction Treatment Center (UMATC) at 1001 W Pratt Street for at least 3 months. The 3-month requirement will help to ensure that patients who enroll in this study have been stabilized on methadone and buprenorphine, which are first-line, evidence-based treatments for OUD.

All procedures associated with this study will be conducted at the UMATC. After completion of brief pre-screen questions to determine eligibility (i.e., age, tobacco use status, and plans to quit smoking), patients will complete a baseline session (BL) and follow-up visits at weeks 2, 6, and 8 lasting between 30-90 minutes each with a total time of participation in the study of approximately 3-4 hours. Each session will include computerized assessments of tobacco and other substance use, health status, mood, and functioning. In addition, patients will be asked to provide a sample of their breath by breathing into a handheld device that measures air breath carbon monoxide levels.

At baseline, participants will be randomly assigned using a number generator to one of two conditions during the baseline session.

1) standard, brief advice for motivating patients to quit (including linkage to a smoking cessation phone quitline) or 2) education on tobacco harms and provisions of NJOY Ace e-cigarette (menthol or tobacco flavor depending on patient preference). NJOY Ace e-cigarettes are a consumer product that has been authorized by the United States Food and Drug Administration. Participants will also be given disposable pods prefilled with nicotine. When the pod is empty, the participant will throw it away and replace it with a new pod provided by the study staff. Participants will be asked to use as little or as much of the e-cigarette during their study participation, including choosing not to use the product.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years or older; currently in treatment for opioid use disorder for at least 3 months
2. currently use tobacco (>100 cigarettes in lifetime and smoke every day or some days)
3. xpired air CO >8ppm
4. does not regularly use e-cigarettes (regular use defined as use in the past month for 2 or more consecutive days)
5. not pregnant or breastfeeding

Exclusion Criteria:

1. individuals trying to stop smoking or have a plan to quit smoking
2. people age 49 or younger
3. people who do not currently smoke tobacco

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Intention to quit smoking in next month | up to 8 weeks
  Measured by self-report in response to following question "Do you intend to stop smoking in the next month?"
Change in cigarettes smoked per day (percent change) | up to 8 weeks
  Measured by self-report during study sessions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Addiction Treatment Center (UMATC), Baltimore, Maryland, United States